CLINICAL TRIAL: NCT01099566
Title: The Role of the P2Y12 Receptor in Tissue Factor Induced Coagulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Bernd Jilma, MD, Medical University of Vienna, Department of Clinical Pharmacology
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPSP2Y12; 2008-001320-32 (EudraCT Number)
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Healthy Volunteers; Sepsis
Keywords: human endotoxemia; tissue factor induced coagulation; platelet activation; thienopyridines
MeSH Terms: conditions — Sepsis | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Experimental)
  Interventions: Drug: Prasugrel
- pills consisting of lactose-starch (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prasugrel — Prasugrel will be given as loading dose (60mg) on the first trial day two hours prior to endotoxin infusion. Prasugrel is an orally administered prodrug that is converted in the liver by CYP to its active metabolite.
  Other Names: Generic name: Prasugrel; Brand name: Efient; Manufacturer: Eli Lilly; Dose: 60mg loading dose (6 tablets a 10mg) on trial day 1
  Arms: Prasugrel
Drug: Placebo — A pharmacist not otherwise involved in the trial will encapsulate pills consisting of lactose-starch. Six pills will be administered as placebo 2 hours before LPS administration on trial day 1.
  Other Names: Content: Pills consisting of lactose-starch; Manufacturer: AKH Anstaltsapotheke; Dose: Same number of pills as in the prasugrel period (6 tablets on trial day 1); identically encapsulated by a pharmacist not otherwise involved in the trial
  Arms: pills consisting of lactose-starch

SUMMARY:
Severe sepsis still carries a high mortality rate despite advantages in intensive care medicine and antimicrobial therapy. The inflammatory and procoagulant host response to infection are intricately linked and interactions between platelets, leukocytes and the endothelium play a central role in the pathogenesis of septic shock and disseminated intravascular coagulation (DIC). Interestingly, one key player cell in coagulation, i.e. the platelet, has been somewhat neglected as to its position in the pathogenesis of coagulation abnormalities in sepsis. However, thienopyridines, irreversible platelet P2Y12 ADP-receptor antagonists, e.g. prasugrel, could potentially provide beneficial anticoagulatory and antiinflammatory effects: P2Y12 ADP-receptor antagonists reduce TF-induced coagulation activation in various ex vivo and in vitro models. Moreover, various lines of evidence indicate that thienopyridines may block platelet leukocyte interactions and thereby reduce the propagation of the coagulation and inflammation process.

LPS-infusion in healthy volunteers provides a standardized model to safely study non overt DIC and to document possible effects of therapeutic and prophylactic interventions.

The investigators hypothesize that thienopyridines, irreversible platelet P2Y12 ADP-receptor antagonists, may blunt TF-triggered coagulation activation in humans, which will be studied in a TF-dependent coagulation model in humans.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities.
* Men aged >18 and <41 years
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Known or suspected allergy to trial product or related products (Prasugrel, Clopidogrel, Ticlopidine)
* Known or suspected hereditary problems of galactose intolerance, Lapp lactase deficiency or glucosegalactose malabsorption
* Treatment with an investigational drug within three weeks prior to this trial
* Treatment with a drug (e.g. ketoconazole, omeprazole) that interferes with cytochrome P450, the enzyme responsible for the conversion of prasugrel to its active form, three weeks prior to this trial
* Participation in an LPS trial within the last 6 weeks
* Smoking of more than 5 cigarettes per day
* Hereditary deficiency of protein C or S, or a mutation of FV (Leiden), or any other known abnormality affecting coagulation, fibrinolysis or platelet function
* History of gastro-duodenal ulcera, cardiovascular disease, vasculitis, diabetes mellitus, or hypertension
* History of brain tumor or history of neurosurgery
* Hemorrhagic diathesis, trauma or surgery within last 3 months
* History of hemorrhagic retinopathy
* Hematuria or detection of occult blood in stool sample
* Liver or kidney dysfunction
* Regular use of medication or abuse of alcohol
* Use of any medication within one week prior to the first trial day
* Symptoms of a clinically relevant illness in the 3 weeks before the first trial day
* Excessive sporting activities
* Weight >95kg and <60kg

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
prothrombin fragments (F1+2) | -2 to 24 hours after LPS infusion
  To explore whether P2Y12 ADP-receptor antagonism can block activation of the coagulation cascade induced by endotoxemia, in particular decrease LPS mediated thrombin formation as measured by prothrombin fragment (F1+2).

SECONDARY OUTCOMES:
platelet-leukocyte co-aggregation | -2 to 24 hours after LPS infusion
  to explore whether P2Y12 ADP-receptor antagonism decreases platelet -leukocyte co-aggregation
tissue factor expression | -2 to 24 hours after LPS infusion
  to investigate the influence of P2Y12 ADP-receptor antagonism on tissue factor expression
anti-platelet effects of prasugrel | -2 to 24 hours after LPS infusion
  to explore if low dose endotoxemia interferes with the anti-platelet effects of prasugrel

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Background] Jilma B, Blann A, Pernerstorfer T, Stohlawetz P, Eichler HG, Vondrovec B, Amiral J, Richter V, Wagner OF. Regulation of adhesion molecules during human endotoxemia. No acute effects of aspirin. Am J Respir Crit Care Med. 1999 Mar;159(3):857-63. doi: 10.1164/ajrccm.159.3.9805087. PMID 10051263
- [Background] Pernerstorfer T, Hollenstein U, Hansen JB, Stohlawetz P, Eichler HG, Handler S, Speiser W, Jilma B. Lepirudin blunts endotoxin-induced coagulation activation. Blood. 2000 Mar 1;95(5):1729-34. PMID 10688831
- [Background] Mavrommatis AC, Theodoridis T, Orfanidou A, Roussos C, Christopoulou-Kokkinou V, Zakynthinos S. Coagulation system and platelets are fully activated in uncomplicated sepsis. Crit Care Med. 2000 Feb;28(2):451-7. doi: 10.1097/00003246-200002000-00027. PMID 10708182
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Kirschenbaum LA, Aziz M, Astiz ME, Saha DC, Rackow EC. Influence of rheologic changes and platelet-neutrophil interactions on cell filtration in sepsis. Am J Respir Crit Care Med. 2000 May;161(5):1602-7. doi: 10.1164/ajrccm.161.5.9902105. PMID 10806162
- [Derived] Spiel AO, Derhaschnig U, Schwameis M, Bartko J, Siller-Matula JM, Jilma B. Effects of prasugrel on platelet inhibition during systemic endotoxaemia: a randomized controlled trial. Clin Sci (Lond). 2012 Nov;123(10):591-600. doi: 10.1042/CS20120194. PMID 22646240